CLINICAL TRIAL: NCT01567774
Title: Pharmacodynamic Effects of Atorvastatin vs. Rosuvastatin on pLatelet Reactivity in Stable Patients With Coronary Artery Disease Treated With Dual Antiplatelet Therapy
Brief Title: Pharmacodynamic Effects of Atorvastatin vs. Rosuvastatin on Platelet Reactivity
Acronym: PEARL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 198/2012/D
Record Dates: First submitted 2012-03-29; First posted 2012-03-30 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; dual antiplatelet therapy; atorvastatin; rosuvastatin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): Patients will receive randomly atorvastatin (20 mg day) for 30 days
  Interventions: Drug: Atorvastatin
- Rosuvastatin (Active Comparator): Patients will receive randomly rosuvastatin (10 mg per day) for 30 days
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Atorvastatin — os, 20 mg, once per day, for 30 days
  Other Names: Norvasc, Pfizer, USA
  Arms: Atorvastatin
Drug: Rosuvastatin — os, 10 mg, once per day, for 30 days
  Other Names: Crestor, AstraZeneca, UK
  Arms: Rosuvastatin

SUMMARY:
Patients with coronary artery disease (CAD) are often treated with dual antiplatelet therapy (DAT), including aspirin and clopidogrel, to prevent from recurrent atherothrombotic events.

Levels of platelet reactivity in patients on DAT can be influenced by concomitant treatment with medications that inhibit the CYP3A4 system involved in the activation of clopidogrel.

Atorvastatin and simvastatin are metabolized by CYP3A4 [Clin pharmacokinetic 2002; 41: 343-70], whereas the cytochrome P450 mediated metabolism of rosuvastatin appears to be minimal and principally mediated by the 2C9 isoenzyme, with little involvement of CYP3A4 [Clin Ther 2003; 25: 2822-5.].

Previous studies comparing atorvastatin versus rosuvastatin by means of ex vivo platelet function tests have yielded conflicting results.

DETAILED DESCRIPTION:
At least 1 month after starting DAT (clopidogrel 75 mg and aspirin 100 mg), patients will receive randomly atorvastatin (20 mg day, N=50) or rosuvastatin (10 mg bid, N=50) for 30 days (until T-1).

At this time-point, there will be a wash-out period of 15 days after the first treatment with atorvastatin or rosuvastatin in order to avoid any carry-over effect.

Afterwards, a cross-over will be performed, and patients will be switched to the other drug which will be continued for further 30 days (until T-2).

ELIGIBILITY:
Inclusion Criteria:

* Angiographically-proven coronary artery disease
* Class I indication to DAT because of recent (<12 months) percutaneous coronary intervention and/or recent acute coronary syndrome (<12 months)
* Stable clinical conditions
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

* Use of other drug interfering with CYP activity such as proton pump inhibitors
* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units | After 30 days of treatment with each drug
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California])

SECONDARY OUTCOMES:
Frequency of high platelet reactivity | After 30 days of treatment with each drug
  Frequency of high platelet reactivity with the 2 study treatments (as defined by a Platelet Reaction Unit value>240

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — University Sapienza
Locations (2):
- Italy (2):
  - Sapienza University, Rome
  - University Sapienza, Rome

REFERENCES:
- [Derived] Pelliccia F, Rosano G, Marazzi G, Vitale C, Spoletini I, Franzoni F, Speziale G, Polacco M, Greco C, Gaudio C. Pharmacodynamic effects of atorvastatin versus rosuvastatin in coronary artery disease patients with normal platelet reactivity while on dual antiplatelet therapy--the PEARL randomized cross-over study. Eur J Pharmacol. 2014 Feb 15;725:18-22. doi: 10.1016/j.ejphar.2014.01.006. Epub 2014 Jan 17. PMID 24444439